CLINICAL TRIAL: NCT00964834
Title: A Phase I, Single Blind, Randomized, Placebo Controlled, Drug Interaction Study of Intravenous (IV) Valortim® and Intravenous (IV) Doxycycline in Healthy Normal Subjects
Brief Title: Ph1 Study of Valortim and Doxycycline in Humans
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sister trial has SAE investigation underway - sponsor elected to withdraw as study expected to be repeated later
Sponsor: PharmAthene, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Medarex (Industry); Quintiles, Inc. (Industry); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Valerie Riddle, M.D., Vice President and Medical Director, PharmAthene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #0036-08-06; NIAID #08-0054
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax | interventions — Doxycycline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Doxycycline and Valortim (Experimental): Randomized such that sixteen volunteer subjects to be renadomized to receive Doxycycline and Valortim
  Interventions: Drug: Doxycycline and Valortim
- Placebo Antibiotic and Valortim (Experimental): Randomized such that four volunteer subjects to receive Placebo Antibiotic and Valortim.
  Interventions: Drug: Placebo Antibiotic and Valortim
- Placebo Antibiotic and Placebo Valortim (Experimental): Randomized such that four volunteer subjects to receive Placebo Antibiotic and Placebo Valortim.
  Interventions: Drug: Placebo Antibiotic and Placebo Valortim

INTERVENTIONS:
Drug: Doxycycline and Valortim — Days 1-5 100mg IV Doxycycline BID over 60 minutes. Day 6 20mg/kg Valortim IV over 60 minutes.
  Other Names: MDX-1303
  Arms: Doxycycline and Valortim
Drug: Placebo Antibiotic and Valortim — Days 1-5 20mg/kg IV Normal Saline BID over 60 minutes. Day 6 20mg/kg IV Valortim over 60 minutes.
  Other Names: MDX-1303
  Arms: Placebo Antibiotic and Valortim
Drug: Placebo Antibiotic and Placebo Valortim — Days 1-5 200mL IV Normal Saline for Placebo Antibiotic BID over 60 minutes. Day 6 20mg/kg IV Normal Saline for Placebo Valortim over 60 minutes.
  Other Names: Saline
  Arms: Placebo Antibiotic and Placebo Valortim

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of short-term dosing of IV doxycycline when administered concomitantly with IV Valortim in normal healthy human subjects.

DETAILED DESCRIPTION:
Valortim (MDX-1303) is a fully human monoclonal antibody (hmAb) with a high affinity for Bacillus anthracis protective antigen (PA). Valortim is designed to target PA, which is one of three plasmid-encoded proteins that together form the toxins released by B. anthracis. Individually, these proteins (protective antigen (PA), lethal factor (LF) and edema factor (EF)) are inactive. Toxic effects require the transport of LF and EF into the host cell, mediated by the activity of PA. Valortim binds to PA and interferes with the activity of the toxins. Based on both non-clinical and clinical data, Valortim may have utility for the pre- and post-exposure prophylaxis of individuals exposed to, or at risk of exposure to, B. anthracis and for the treatment of individuals displaying symptoms of inhalational anthrax. Because the treatment of inhalational anthrax includes the use of antibiotics such as tetracyclines, it is necessary to demonstrate that there are no adverse interactions between newer therapeutic interventions and these medications. The purpose of this study is to assess the pharmacokinetics of doxycycline (a commonly used tetracycline for both treatment and post-exposure prophylaxis of anthrax) and Valortim following co-administration, as well as the safety and tolerability of these medications when administered concomitantly. These data are intended to support the use of Valortim as a treatment for inhalational anthrax.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy normal male or female subjects 18 to 65 years of age on Day -1 of the study
2. Subject must have read, understood, and provided written informed consent after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures
3. In the opinion of the Investigator, subjects should be in generally good health, based upon prestudy medical history, physical examination, ECG and laboratory tests (see Appendix H)
4. Laboratory screening values (i.e., hematology, clinical chemistries and urinalysis tests) must be within study-defined ranges (See Appendix G).
5. No detectable antibody to B. anthracis Protective Antigen (PA-IgG) as measured by ELISA testing at study Screening
6. Women of childbearing potential may be enrolled if one of the following criteria applies:

   1. Must be using an effective form of contraception (e.g., oral contraceptives,, IUD, injected or implanted hormonal contraception, double barrier method of condom and spermicide, diaphragm with spermicide or sponge with spermicide) for at least one month prior to study entry, must have maintained a normal menstrual pattern for the three months prior to study entry and have a negative pregnancy test at the time of admission to the unit. Women must be willing to continue this contraception throughout the course of the study.
   2. Is sexually abstinent
   3. Is monogamous with a vasectomized partner (> 3 months prior)
   4. Is postmenopausal (i.e., no cycle for at least the previous 12 months, is of menopausal age (> 45 years) and has a negative urine pregnancy test prior to enrollment into the study and a negative serum pregnancy test on Day -1)
   5. Is surgically sterilized (confirmed by medical record review)
   6. Has had a total hysterectomy a minimum of 3 months prior to dosing on Day 1 (confirmed by medical record review)
7. Sexually active male subjects may be enrolled if one of the following criteria applies:

   1. Has had a vasectomy (> 3 months prior to study entry, confirmed by medical record review)
   2. Using condoms and whose partner is using an acceptable form of contraception (IUD, oral contraceptives, birth control patch or vaginal ring, injectable or implanted contraceptives, or tubal ligation [surgical sterilization]) for the duration of the study
   3. Is sexually abstinent
8. Female subjects must have a negative urine pregnancy test at study Screening and a negative serum pregnancy test on admission to the Phase I unit at Day -1
9. Female subjects using injectable, transdermal, vaginal ring, oral contraceptives, or an IUD must agree to also use a barrier method (i.e. male condom, female condom, diaphragm, cervical cap) for the duration of their participation in the study.
10. Agreement to not receive any vaccinations from Day -1 through to 31 days post Valortim dosing. Vaccination against B. anthracis is prohibited during the study.
11. Body Mass Index (BMI) ≥ 19 and ≤ 30 (see Appendix C)
12. Abstinence from alcohol for 24 hours prior to study drug administration until discharge from the Phase I unit

Exclusion Criteria:

1. Prior known or suspected exposure to B. anthracis
2. Prior vaccination for B. anthracis
3. Any participants in the original FTIH study of Valortim.
4. History of drug or alcohol abuse i.e. having been treated either in an in-patient or out-patient facility within 12 months of study Screening
5. Positive drug result and/or positive alcohol result at time of study Screening or at Day -1
6. Smoke more than 10 cigarettes per day for the last 6 months
7. Treatment with an investigational agent within 30 days or 5 half-lives (whichever is longer) of study Screening
8. Use of systemic immunosuppressive agents within 12 months of study Screening. Individuals who have received prednisone or its equivalent in doses of less than 20 mg/day for 14 days or less, as long as it occurred more than 1 month prior to them entering the study and as long as there is no clinical or laboratory evidence of immunosuppression, may be considered for enrollment
9. Use of laxatives within 24 hours prior to dosing
10. Use of proton pump inhibitors within 72 hours prior to dosing
11. History of asthma requiring any use of inhaled or oral medication within the previous 5 years
12. History of hepatic or renal impairment or diabetes
13. Clinically significant medical or psychiatric condition that, in the opinion of the Investigator, may impair study participation to include ongoing recent illness, new medications prescribed in the previous 6 weeks or use of immunosuppressive agents
14. Electrocardiogram with evidence of clinically significant conduction abnormalities or active ischemia (as determined by the Principal Investigator) at the time of study screening
15. Donation of one or more pints of blood 30 days prior to study Screening visit or donation prior to completion of Day 34 of the study
16. Donation of plasma within 14 days prior to study Screening visit or donation prior to completion of Day 34 of the study
17. Vaccinations within 30 days prior to Day -1 through to 31 days post Valortim dosing on Day 6.
18. Prior known serum positivity for human immunodeficiency virus (HIV) antibodies, hepatitis B (surface antigen) or hepatitis C as determined at study Screening
19. Prior known allergy or allergic reaction to doxycycline or any of the group of antibiotics known as tetracyclines
20. Current treatment with, or use of, anticoagulants, antibiotics, barbiturates and anti-epileptic drugs
21. Diagnosis of photosensitivity, including, but not limited to, a history of phototoxic and/or photoallergic reactions to medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determination of changes from baseline for clinical laboratory tests and urinalysis, blood pressure, heart rate, respiratory rate, body temperature, physical examination and ECG | 137 days

SECONDARY OUTCOMES:
Evaluation of PK parameters for IV administration of doxycycline when dosed concomitantly with Valortim | 137 days

CONTACTS AND LOCATIONS:
Overall Officials: Daivd Mathews, M.D., Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States

REFERENCES:
- See also: Click here for more information about this study. — http://www.StudyForChange.com